CLINICAL TRIAL: NCT05414955
Title: Boom-IBD Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boomerang Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Boom-IBD
Record Dates: First submitted 2022-05-10; First posted 2022-06-10 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: IBD
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treated (Experimental): Patients implanted with neuromodulation
  Interventions: Device: Neuromodulation

INTERVENTIONS:
Device: Neuromodulation — Neuromodulation

SUMMARY:
Feasibility study of neuromodulation in patients with IBD.

DETAILED DESCRIPTION:
The study will evaluate responses of patients with IBD treated with neuromodulation at various intervals.

ELIGIBILITY:
General Inclusion Criteria:

* Male or female
* 18 to 75 years of age
* Diagnosed with Crohn's Disease or ulcerative colitis
* Ability and willingness to consent to participate by signing the informed consent form
* Ability to comply with the protocol and willingness to comply with all follow-up requirements
* Still have part or all of their colon

General Exclusion Criteria (The subject must not meet ANY of the following criteria):

* Any significant medical condition that is likely to interfere with study procedures, device operation, or likely to confound the results of the study
* Any psychiatric or personality disorder at the discretion of the study investigator
* Any active bacterial infection with a risk of bacteremia or sepsis (e.g. presence of abscess)
* Active clostridium difficile infection of the colon
* Active cytomegalovirus (CMV) infection of the colon
* Evidence of colonic perforation
* Fulminant colitis requiring emergency surgery
* Microscopic, ischemic or infectious colitis
* Unresected neoplasia of the colon
* Colonic stricture unable to pass a colonoscope
* History of cancer including melanoma (except for localized skin cancers) within 2 years
* Participation in another clinical trial within the past 30 days of device implant
* Investigational drug for the treatment of inflammatory bowel disease within 6 months of device implant
* Inability to operate the patient programmer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Disease Activity Index | up to 1 year
  CDAI (Crohn's Disease Activity Index Score) or MAYO Score (ulcerative colitis)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Phillip Fleshner, Inc., Los Angeles, California
  - Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - CU Anschutz, Aurora, Colorado
  - Kansas Gastroenterology, Wichita, Kansas
  - Las Vegas Medical Research, Las Vegas, Nevada
  - The Mount Sinai Medical Center, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - University of Pennsylvania, Perelman School of Medicine Division of Colorectal Surgery, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No